CLINICAL TRIAL: NCT06243666
Title: Long-term Effectiveness and Immuno-persistence Study of a Recombinant Human Papillomavirus 16/18 Bivalent Vaccine in Girls Aged 9-17 Years
Brief Title: Long-term Effectiveness and Immuno-persistence Study of a Recombinant HPV 16/18 Bivalent Vaccine in Preadolescent Girls
Status: Active, not recruiting | Type: Observational
Sponsor: Xiamen University (Other)
Collaborators: Xiamen Innovax Biotech Co., Ltd (Industry); Center for Disease Control and Prevention, Sheyang County, Yancheng City, Jiangsu Province, China (Unknown)
Responsible Party: Principal Investigator, Jun Zhang, professor, Xiamen University
Other Study IDs: HPV-PRO-006-4
Record Dates: First submitted 2024-01-29; First posted 2024-02-06 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Cervical Intraepithelial Neoplasia; Cervical Cancer; Persistent Infection
Keywords: Human Papilloma Virus 16; Human Papilloma Virus 18; Adolescent girl; Long-term Effectiveness; Immuno-persistence
MeSH Terms: conditions — Uterine Cervical Dysplasia; Uterine Cervical Neoplasms; Persistent Infection | interventions — Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Vaccine group for long-term effectiveness evaluation: No intervention was implemented in this study. Participants who have participated in the immunobridging clinical trial of the bivalent HPV vaccine (Unique Protocol ID:HPV-PRO-006,Identifiers: NCT02562508) and were aged 9-17 years at the time of enrollment, and have received at least one dose of the vaccine were recruited as the vaccine group for long-term effectiveness evaluation.
  Interventions: Biological: Recombinant Human Papillomavirus Bivalent (Types 16, 18) Vaccine (Escherichia coli)
- Control group for long-term effectiveness evaluation: No intervention was implemented in this study. Participants with no previous HPV vaccination history were recruited as the control group for long-term effectiveness evaluation.
  Interventions: Other: No intervention
- Vaccine group for immuno-persistence evaluation: No intervention was implemented in this study. Participants who have participated in the immunobridging clinical trial of the bivalent HPV vaccine (Unique Protocol ID:HPV-PRO-006,Identifiers: NCT02562508) and were aged 9-26 years at the time of enrollment, and have received at least one dose of the vaccine were recruited as the vaccine group for immuno-persistence evaluation.
  Interventions: Biological: Recombinant Human Papillomavirus Bivalent (Types 16, 18) Vaccine (Escherichia coli)

INTERVENTIONS:
Biological: Recombinant Human Papillomavirus Bivalent (Types 16, 18) Vaccine (Escherichia coli) — The bivalent HPV-16/18 vaccine was a mixture of two aluminum hydroxide adjuvant-absorbed recombinant L1 VLPs of HPV-16 and HPV-18 expressed in E. coli. A 0.5 ml dose of the bivalent HPV test vaccine comprised 40 μg of HPV-16 and 20 μg of HPV-18 L1 VLPs absorbed with 208 μg of aluminum adjuvant.
  Groups: Vaccine group for long-term effectiveness evaluation
Other: No intervention — No intervention was implemented.
  Groups: Control group for long-term effectiveness evaluation
Biological: Recombinant Human Papillomavirus Bivalent (Types 16, 18) Vaccine (Escherichia coli) — The bivalent HPV-16/18 vaccine was a mixture of two aluminum hydroxide adjuvant-absorbed recombinant L1 VLPs of HPV-16 and HPV-18 expressed in E. coli. A 0.5 ml dose of the bivalent HPV test vaccine comprised 40 μg of HPV-16 and 20 μg of HPV-18 L1 VLPs absorbed with 208 μg of aluminum adjuvant.
  Groups: Vaccine group for immuno-persistence evaluation

SUMMARY:
The primary objective of this study is to evaluate the protective efficacy against future infections of HPV types 16/18 or related diseases and immuno-persistence (type specific IgG antibody) of the bivalent HPV vaccine in young female populations aged 9-17 years.

DETAILED DESCRIPTION:
This is a follow-up study that is based on the bridging study of a recombinant human papillomavirus 16/18 bivalent vaccine in preadolescent girls(Unique Protocol ID:HPV-PRO-006,Identifiers: NCT02562508) . This study proposes to conduct a prospective cohort study based on the cohort population from the immunobridging clinical trial of the bivalent HPV vaccine (Unique Protocol ID:HPV-PRO-006,Identifiers: NCT02562508) . By matching control groups according to factors such as age and education level, and through long-term follow-up, this research aims to elucidate the protective efficacy of the bivalent HPV vaccine against future infections of HPV types 16/18/31/33/45 or related diseases in young female populations aged 9-17 years. Additionally, the study will evaluate the persistence of vaccine-induced antibodies, investigate the potential for type replacement/competition phenomena post-vaccination and assess oral HPV infections in the cohort population.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be at least 18 years old;
* Participants who have participated in the immunobridging clinical trial of the bivalent HPV vaccine (Unique Protocol ID:HPV-PRO-006,Identifiers: NCT02562508) and have received at least one dose of the vaccine (only applicable to the vaccine group);
* Able to understand the study procedure and have the ability to comply with the protocol requirements (e.g., collection of biological samples and regular follow-up) and sign a written informed consent form;

Exclusion Criteria:

* Participants who did not experience sexual debut;*
* Participants with acute cervical inflammation and acute lower genital tract infection;*
* Participants during menstruation, or have vaginal medication, sexual behavior within two days (48 hours) before the visit, which may affect gynecological examinations and specimens collection;*
* Participants in the vaccine group have used other HPV vaccine products (including both marketed and unmarketed vaccines) after participating in the immunobridging clinical trial of the bivalent HPV vaccine (Unique Protocol ID: HPV-PRO-006, Identifiers: NCT02562508); Participants in the control group have used HPV vaccine products (including both marketed and unmarketed vaccines);
* According to the judgement of investigator, various medical, psychological, social, vocational or other factors that are not suitable for participating in the study.

  * Note: For criteria marked with an asterisk (*), if the participant meets that exclusion criterion, it does not affect the blood sample collection.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants who participated in the bridging study (Unique Protocol ID: HPV-PRO-006, Identifiers: NCT02562508) and received at least one dose will be recruited as vaccine group. Participants with no previous HPV vaccination history were recruited as the control group.
Sampling Method: Non-Probability Sample
Enrollment: 2188 (Estimated)
Dates: Start 2024-02-20 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of persistent infection, transient infection, and cervical precancerous CIN1+ lesions associated with HPV types 16 and 18 | 8-10 years after the first dose
  To evaluate the efficacy of the bivalent vaccine against this outcome
Anti-HPV 16 and 18 IgG antibody seropositive rates and geometric mean concentrations | 9 years after the first dose
  To detect the anti-HPV 16 and anti-HPV 18 type-specific IgG antibody level 9 years after the first dose

SECONDARY OUTCOMES:
Incidence of persistent infection, transient infection, and cervical precancerous CIN1+ lesions associated with HPV types 31/33/45 | 8-10 years after the first dose
  To evaluate the efficacy of the bivalent vaccine against this outcome

OTHER OUTCOMES:
Incidence of persistent infections, transient infections, and CIN1+ lesions associated with other high-risk types (except HPV types 16, 18, 31, 33, and 45). | 8-10 years after the first dose
  To investigate the potential for type replacement/competition phenomena post-vaccination
Incidence of transient and persistent infections with oral HPV | 8-10 years after the first dose
  To explore the incidence of transient and persistent oral HPV infections in vaccinated and unvaccinated populations

CONTACTS AND LOCATIONS:
Overall Officials: Ting Wu, Ph. D., Principal Investigator — Xiamen University; Jun Zhang, MSc, Study Chair — Xiamen University
Locations (1):
- Sheyang County Center for Disease Control and Prevention, Yancheng, Jiangsu, China